CLINICAL TRIAL: NCT03886753
Title: Pharmacokinetic and Pharmacodynamic Study of Ilera Medical Marijuana Products
Brief Title: Pharmacokinetic (PK) and Pharmacodynamics (PD) Study of Ilera Specific Products
Acronym: Ilera
Status: Terminated | Type: Observational
Why Stopped: Feasibility
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Ilera Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18-015787
Record Dates: First submitted 2019-01-14; First posted 2019-03-22 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: ALS; Autism Spectrum Disorder; Cancer; Spasticity, Muscle; Dyskinetic Syndrome; Epilepsy; Glaucoma; Huntington Disease; Inflammatory Bowel Disease (IBD); Multiple Sclerosis; Neuropathy; Opioid Use; Parkinson Disease; HIV/AIDS; Ptsd; Intractable Pain; Sickle Cell Disease; Terminal Illness
MeSH Terms: conditions — Autism Spectrum Disorder; Neoplasms; Muscle Spasticity; Dyskinesias; Epilepsy; Glaucoma; Huntington Disease; Inflammatory Bowel Diseases; Multiple Sclerosis; Parkinson Disease; Acquired Immunodeficiency Syndrome; Stress Disorders, Post-Traumatic; Pain, Intractable; Anemia, Sickle Cell | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will ask patients if we can retain their specimens for future studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Ease: Subjects using Ease as standard treatment. Registry and PK sampling
  Interventions: Other: Registry; Other: PK microsampling of blood
- Dream: Subjects using Dream as standard treatment. Registry and PK sampling
  Interventions: Other: Registry; Other: PK microsampling of blood
- Soothe: Subjects using Soothe as standard treatment. Registry and PK sampling
  Interventions: Other: Registry; Other: PK microsampling of blood
- Shine: Those subjects using Shine as standard treatment. Registry and PK sampling
  Interventions: Other: Registry; Other: PK microsampling of blood

INTERVENTIONS:
Other: Registry — Collect data on subjects
Other: PK microsampling of blood — Obtain 5 microsamples of blood from subjects via a fingerstick.

SUMMARY:
This is an observational study of medical marijuana manufactured and dispensed by Ilera and given as standard treatment for a variety of approved serious medical conditions as defined by individual state law. All patients who are receiving one of the four formulations (Dream, Soothe, Shine and Ease) of medical marijuana will be provided a study flyer and asked to contact the study team via phone or email. Once the study team confirms eligibility, the study team will meet the subject face-to-face most likely at their dispensary (or other mutually agreeable location) and obtain informed consent, and assent when appropriate. Initial baseline demographic information, medical history and medication inventory will be completed. Also, since it is possible that the Investigators will enroll subjects across the region, Investigators anticipate the need to seek consent over the phone for many patients. This will be done via Skype, Go to Meeting, Facetime or similar platforms so that the Investigators can have a face to face interaction with the potential subjects. Regardless of where this discussion takes place (i.e., in person or via the web), all reasonable safeguards to ensure patient privacy will be taken. Patients or their legally authorized representative (LAR) will be given sufficient (i.e., up to several hours/days) to make a decision to participate in this study. Study staff will fax or email the consent form for their signature and no study procedures will begin until the signed consent form is received by the study team. The subjects or their LARs will be instructed on obtaining the blood samples. Blood draws will be completed in the subjects' home after one of their standard doses is taken.

DETAILED DESCRIPTION:
This is a prospective PK/PD study that will include patients who are currently legally consuming one of the four medical marijuana formulations (Dream, Soothe, Shine and Ease) from Ilera Healthcare as part of their standard therapy for one of the state approved serious medical conditions.

Part 1 of the study consists of intake data of select subjects.

* The patients will be identified at a dispensary that offers Ilera products.
* Patients be given a flyer about the study by either study staff or dispensary staff.
* Eligible patients will be asked to contact the study team if they are interested in the study.
* If the patient is interested, a face-to-face (in person at the dispensary or in the patients home or other agreed upon location) consent/assent will be obtained.
* Also, since it is possible that Investigators will enroll subjects across the region, Investigators anticipate the need to seek consent over the phone for many patients. This will be done via Skype, Go to Meeting, Facetime or similar platforms so that the investigators can have a face to face interaction with the potential subjects. Investigators will obtain written consent in all cases. Investigators will have them sign and fax or email/scan the signed consent form back to the study team.
* Once consent is obtained demographic information will be collected as well as a medical and medication history and several questions related specifically to the medical marijuana product and its perceived effectiveness.
* The data will be recorded in the REDCAP database. Part 2 of the study consists of pharmacokinetic evaluation of select subjects.
* Parents/ care providers/ patients when appropriate will undergo education regarding PK sample acquisition
* PK blood samples will be obtained and sent to the Children's Hospital of Philadelphia (CHOP) for determination of cannibidiol/ Tetrahydrocannabinol/ cannabinol (CBD/THC/CBN) concentrations
* PK and PD analysis will occur

ELIGIBILITY:
Inclusion Criteria:

* Individuals who consume either Dream, Shine, Soothe or Ease medical marijuana manufactured by Ilera Heath care in a state which has legalized medical marijuana for state specified serious medical conditions.
* Written informed consent and assent (if applicable)
* Patients greater than 2 years of age

Exclusion Criteria:

* Consumption of marijuana products that are not obtained from a state licensed dispensary
* Non English speaking individuals
* Have consumed a CBD/THC containing product other than the product under study within the 7 days prior to the PK study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 2 years old who are being treated with Dream, Shine, Ease or Soothe products manufactured by Ilera Healthcare for a state approved qualifying medical condition under the PA State Medical Marijuana Program.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in symptoms | 1 year
  Relief of primary indication (perceived therapeutic benefit of product)as reported by parent or caregiver on a 1-10 Lichert scale with 1 being minimally effective and 10 being extremely effective

SECONDARY OUTCOMES:
Description and incidence of patient or caregiver reported side effects | 1 year
  There is no particular instrument used in collecting this data. It is an open ended question where by patients and caregivers report possible side effects from the medical marijuana. Investigators will report the incidence in percentages.
Changes in drug concentrations | 2 years
  The amount of a drug in a given volume of blood plasma, measured as the number of micrograms per milliliter
Rate of bioavailabilty | 2 years
  The degree and rate at which the medication is absorbed by the body's circulatory system, the systemic circulation.
Volume of distribution | 2 years
  The volume of medication that would be necessary to contain the total amount of the administered drug at the same concentration that it is observed in the blood plasma.
Report area under the plasma concentration versus time curve (AUC) | 2 years
  The area under the curve (AUC) is the definite integral in a plot of drug concentration in blood plasma vs. time
Report half-life | 2 years
  Half life is described as how long it takes for half of the dose to be metabolized and eliminated from the bloodstream.
Assess therapeutic range | 2 years
  Comparison of the amount of a therapeutic agent that causes the therapeutic effect to the amount that causes toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Athena F Zuppa, MD MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No